CLINICAL TRIAL: NCT03720964
Title: Mitochondrial Genetics of Presbycusis
Acronym: MITOPRES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC18_0148
Record Dates: First submitted 2018-10-24; First posted 2018-10-26 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Presbycusis; Age Related Hearing Loss
MeSH Terms: conditions — Presbycusis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extracted from blood and urine will be stored in "Centre de Ressources Biologiques" as planed in biocollections "maladies mitochondriales" and "volontaires sains"
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- presbycusis affected patients: affected by a more severe age related hearing loss than expected according to the norm ISO 7029
- controls: not affected by age related hearing loss according to the norm ISO 7029

SUMMARY:
The main goal of this study is to identify mitochondrial mutations associated with presbycusis. Patients affected by severe presbycusis and normal hearing controls (according to ISO7029 norm) will be enrolled if satisfying inclusion criteria (aged from 40 to 80 years old) in existing biocollections in the University Hospital of Angers. After DNA extraction, the mitochondrial genome will be sequenced and data in silico analysed.

DETAILED DESCRIPTION:
The study will be proposed to patients consulting in the ENT department of the University Hospital of Angers. After clinical examination and audiometry recording, the eligibility criteria will be checked and inclusion in biocollections proposed. Presbycusis affected subjects will be enrolled in "Mitochondrial Disease biocollection" and normal hearing controls in "Healthy Volunteer biocollection". These biocollections have been approved by the board comitee "Centre de Protection des Personnes".

After DNA extraction and mitochondrial sequencing, candidate variants will be selected by in silico analysis. The presence of mitochondrial variants in both groups (presbycusis and control) will be compared in multivariate analysis if needed.

The nuclear DNA may be sequenced in order to complete the previous analysis and look for any candidate variant .

ELIGIBILITY:
Inclusion Criteria:

* age related hearing loss more severe than the predicted hearing thresholds according to the norm ISO7029, for the presbycusis population;
* normal hearing according to norm ISO7029 for the control population

Exclusion Criteria:

* deafness diagnosed before 40 years old
* exclusion criteria of one of the biocollection

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is proposed to patients consulting for hearing evaluation in ENT department of University Hospital of Angers.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
identification of mitochondrial mutations associated with presbycusis | the analysis will be conducted at the end of the inclusion of the 200 patients
  Enrichment analysis will be perfomed with CHI2 test after Benjamini correction.

SECONDARY OUTCOMES:
identification of genomic variants associated with presbycusis | the analysis will be conducted at the end of the inclusion of the 200 patients
  enrichment of genomic variants will be analysed
identification of DNA variants associated with environmental susceptibility | the analysis will be conducted at the end of the inclusion of the 200 patients
  subgroup analysis will be performed in accordance with environmental exposition

OTHER OUTCOMES:
identification of clinical features predicting some presbycusis forms | the analysis will be conducted at the end of the inclusion of the 200 patients
  analysis of audiometric data after genetic analysis will be performed

CONTACTS AND LOCATIONS:
Locations (1):
- UH Angers, Angers, France